CLINICAL TRIAL: NCT06525532
Title: Clinical-MRI Evaluation in Patients Undergoing Subtalar Arthrorisis With Resorbable PLLA Endothesis Implant: Prospective Observational Study at 5 Years of Minimum Follow-up
Brief Title: Clinical-MRI Evaluation in Patients Undergoing Subtalar Arthrorisis With Reabsorbable Endorthesis Implant in PLLA
Acronym: CS-RM
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: CS-RM
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Lower Limb Deformity
Keywords: arthrorrhesis; reabsorbable endorthotic implant; subtalar joint; pediatric joint implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: subjects who have undergone surgery for subtalar arthroritis with a reabsorbable endorthotic PLLA implant
  Interventions: Other: follow up

INTERVENTIONS:
Other: follow up — performing a 3 Tesla MRI of the operated foot

SUMMARY:
From the archives of the IRCCS Rizzoli Orthopedic Institute, all cases of arthrorrhesis of the subtalar joint with a reabsorbable endorthotic implant in PLLA will be retrieved. An overall electronic database will be created and all medical records of these cases will be reviewed.

The eligibility of each individual patient will be assessed on the basis of the exclusion and inclusion criteria (non-probability convenience sampling).

The study will not present a control group or comparison groups between therapeutic procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 15 years at the time of surgery
* Arthrorrhosis of the subtalar with reabsorbable endorthotic implant in PLLA
* Minimum follow-up of 5 years

Exclusion Criteria:

* Revisions/explantation of the endorthesis device
* Patients with active acute or chronic infections
* Patients with chronic inflammatory joint diseases
* Patients with previous significant trauma of the lower limbs following surgery
* Patients with pre-existing anomalies of ambulatory kinematics (amputations, neuro-muscular diseases, poliomyelitis, hip dysplasias)
* Patients with cognitive deficits
* - Patients with concomitant neurological pathologies
* Patients suffering from tumor pathology
* Patients with cardiac pacemakers or other prostheses equipped with electronic circuits
* Patients with intracranial metal implants, metal heart valves, vascular clips, ferromagnetic endovascular filters/stents/coils, Swan-Ganz catheters or in any case positioned close to vital anatomical structures
* Patients with orthopedic metal prostheses
* Patients with cochlear implants or fixed hearing aids, lens prostheses with ferromagnetic intra-ocular points, IUD (coil) or splinters made of ferromagnetic material
* Pregnant patients
* Patients with insulin pumps and non-removable contact lenses

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric population with subtalar arthrorisis surgery with reabsorbable endorthesis implant in PLLA
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Instrumental evaluation | At baseline (Day 0)
  Instrumental evaluation with 3 Tesla MRI of the degradation and possible resorption of the implant
evaluation of screw resorption | at baseline
  Clinical and Magnetic Resonance Imaging Results - PMC (nih.gov), Poly-L-lactic acid - hydroxyapatite (PLLA-HA) bioabsorbable interference screws for tibial graft fixation in anterior cruciate ligament (ACL) reconstruction surgery

SECONDARY OUTCOMES:
clinical evaluation - Ankle-Hindfoot score | at baseline (day 0)
  AOFAS: this questionnaire consists of points assigned to nine items divided into three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) for a total of 100 points, the extreme of which represents a normal foot complex -ankle
Quality of life - SF-12 | at baseline
  The SF-12 health questionnaire is a standardized generic instrument for the rapid, economical and disease-free acquisition of the patient's health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Benedetti MG, Ceccarelli F, Berti L, Luciani D, Catani F, Boschi M, Giannini S. Diagnosis of flexible flatfoot in children: a systematic clinical approach. Orthopedics. 2011 Jan 1;34(2):94. doi: 10.3928/01477447-20101221-04. PMID 21323297
- [Result] Kim MK, Lee YS. Kinematic analysis of the lower extremities of subjects with flat feet at different gait speeds. J Phys Ther Sci. 2013 May;25(5):531-3. doi: 10.1589/jpts.25.531. Epub 2013 Jun 29. PMID 24259795